CLINICAL TRIAL: NCT03384979
Title: Randomized Controlled Trial of Optimization of Contrast Agent Dose in CT With Lean Body Weight
Brief Title: Optimization of Contrast Agent Dose in CT With Lean Body Weight
Acronym: CA_LBW
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Head of Radiology, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: LBW_02
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Contrast Agent With Lean Body Weight
MeSH Terms: interventions — Iopamidol

STUDY DESIGN:
Intervention Model Description: The study design is monocentric, comparative, randomized, double blinded. Patients will undergo a CT scan of abdomen (multi-phasic) with contrast agent and will be measured: TBW, height, LBW and body mass index (BMI) through formulas known in literature and with a balance for bioelectrical impedance analysis. There is no administration of drugs other than indicated in the request of the treating physician.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be assigned to the TBW or LBW group based on a randomization generated by a computer, the progressive sequences containing the randomization code will be perform by an outside operator to the experiment group. Only CT technician and nurse that will record patient's data and results from scale analysis will know and will register in which group the patients will be assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TBW protocol (Placebo Comparator): Patients will receive a contrast agent dose based on their TBW as a standard clinic protocol.
  Interventions: Drug: Iopamidol
- LBW protocol (Experimental): Patients will receive a contrast agent dose based on their calculated LBW.
  Interventions: Drug: Iopamidol

INTERVENTIONS:
Drug: Iopamidol — Contrast agent will be adrministered intravenously using total body weight or lean body weight, calculated with bioelectrical impedance analysis balance.
  Other Names: Iomeprolo

SUMMARY:
This study evaluates the different enhancement using a contrast agent dose in computed tomography based on total body weight or based on lean body weight. Half of participants will receive contrast agent dose based on their total body weight, while the other half will receive a dose based on their lean body weight. Our hypothesis is that if contrast agent is administered not basing on total body weight but on lean body weight it is possible to obtain equal or better quality of enhanced images, a reduction of the variability of contrast enhancement, and also a dose reduction in some patients (overweight ones).

DETAILED DESCRIPTION:
Patients will undergo a CT scan of abdomen (multi-phasic) with contrast agent and will be measured: total body weight (TBW), height, lean body weight (LBW) and body mass index (BMI) through formulas known in literature and with a balance for bioelectrical impedance analysis. There is no administration of drugs other than those indicated in the request of the treating physician.

Contrast agent dose:

IOPAMIRO® (Iopamidol) is an x-ray contrast medium of the new generation of non-ionic compounds, which are watersoluble because the molecular structure incorporates hydrophilic groups. Recommended dosage (ml) is 0.5-2.0/kg. Single injection volume depends on the vascular area to be examined.

IOMERON® (Iomeprolo) is an x-ray contrast medium of the new generation of non-ionic compounds, which are watersoluble because the molecular structure incorporates hydrophilic groups. Recommended dosage (ml) is 0.5-2.0/kg. Single injection volume depends on the vascular area to be examined.

Patients will be randomly assigned to undergo one of the two contrast agent protocols.

Control group (TBW protocol): patients will receive a contrast agent dose based on their TBW as a standard clinic protocol with a dose of 0.40 gI/kg of TBW. There are no differences compared to clinical practice.

Experimental group (LBW protocol): patients will receive a contrast agent dose based on their calculated LBW to test our hypothesis with a dose of 0.65 gI/kg of LBW, derived from our pilot study (LBW_01 approved 10/11/2016, registration number 160/int/2016).

If radiologists prefer a more enhanced examination, only scanning with contrast agent will be repeated with the standard dose as the standard clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age;
* Patients who will perform a contrast-enhanced abdominal CT multi-phasic in our institutions;
* Patients able to give informed consent.

Exclusion Criteria:

* history of chronic underlying liver disease (cirrhosis, fatty infiltration of the liver, or glycogen storage disease);
* history of chronic underlying heart disease (congestive heart failure, prior cardiac valve replacement, restrictive and/or constrictive pericarditis);
* multiple myeloma;
* hypersensitivity to iodine-containing compounds;
* renal insufficiency (serum creatinine level ≤ 1.8 mg/dL [159.12 µmol/L]) or patients with renal failure (eGR <30 ml/min/1.73 m2);
* patients with antecubital vein that, at medical evaluation, cannot sustain the flow rate of CA injection (see below);
* patients carrier of prosthesis or metal bullets, pacemaker or stimulators;
* patients with liver diseases that affect the entire parenchyma;
* fragile patients which, after radiologist evaluation, require lower dose of CA;
* pregnancy;
* general contraindications to CT examination or reasoned decision of the radiologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Contrast Enhancement | 1 day
  The liver contrast enhancement (ΔCEL) will be calculated as the difference between the CT value measured in the venous phase and that measured before contrast injection.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No